CLINICAL TRIAL: NCT04105569
Title: An Atlas of Experimental Gingivitis in Humans at Single Cell Resolution
Brief Title: Atlas of Experimental Gingivitis in Humans
Acronym: ATL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Sunstar, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-0183
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Enrolled subjects will be included in an experimental gingivitis model (SIBO) for 21 days and use an acrylic stent fabricated before and dispensed at the baseline appointment
  Interventions: Procedure: Stent-Induced Biofilm Overgrowth

INTERVENTIONS:
Procedure: Stent-Induced Biofilm Overgrowth — Customized acrylic dental (sextant) stent will be used during brushing for 21 days to influence reversible gingival tissue inflammation.
  Other Names: Dental Stent

SUMMARY:
Pilot case series with a split-mouth design to track subjects with known exposure (dental biofilm accumulation) over 21 days. Descriptive design, using single cell RNA sequencing as a "digital biopsy" to catalog and contrast inflamed versus non-inflamed tissues from within the same mouth and across patients. Specimens (human) will biobanked from the 'digital biopsy' site for future analysis, including: Gingival crevicular fluid, oral epithelial stem/progenitor cells, and plaque samples, for 'omics analyses including metabolomics, microbiomic, and genomic data.

DETAILED DESCRIPTION:
Purpose is to conduct the first study of human gingiva in health and after biofilm-induced inflammation in the gingiva using scRNAseq. The pilot will involve induction of experimental gingivitis in all participants.

Participants include recruitment of 6 participants. Following consenting, screening, and enrollment, a customized acrylic stent will be used only on the selected sextant/teeth specified in the protocol, and only during tooth brushing to prevent oral hygiene in selected sextant/teeth. After the completion of the 3-week gingivitis induction phase, participants will enter a 2 week resolution phase. In the resolution phase, participants will reinstate full mouth oral hygiene, with the exception of flossing. Oral prophylaxis will be performed to regain health. During the 3 week gingivitis induction phase, participants will be required to return to the clinic every 7 days for safety checks.

Study Procedures (methods): Medical history, demographics (height/weight), urine based pregnancy test, vital signs (to include blood pressures, and pulse), standard dental clinical measures (to include plaque index, gingival index, bleeding on probing, and clinical attachment level), alginate impressions taken for fabrication of an acrylic stent (mouth guard), 2 gingival biopsies, 4 subgingival (below the gum line) plaque samples, 4 Gingival Crevicular Fluid (naturally occurring fluid between the gum and teeth) samples, and adult prophylaxis

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females between the age of 18 and 30 years.
* Non-diabetic and no history of smoking within the last 5 years.
* Have read, understood and signed an informed consent form.
* Must be able and willing to follow study procedures and instructions.
* Must have at least 3 natural adjacent teeth in both maxillary (top) posterior sextants that will be selected for baseline gingival biopsy and SIBO gingival biopsy.
* Must be in good general health, as evidenced by medical hx (exclusion conditions defined under subject exclusion criteria below).
* Females of childbearing capacity must be willing to have pregnancy test to confirm they are not pregnant.

Exclusion Criteria

* History of intravenous bisphosphonates.
* Current or history (less than 5 years) of tobacco use in any form prior to enrollment (self-report)
* Chronic disease with oral manifestations including diabetes mellitus.
* Infectious disease such as hepatitis, HIV, or tuberculosis.
* Anemia or other blood dyscrasias.
* Currently taking anticoagulant therapy or drugs, such as heparin or warfarin.
* Those requiring antibiotic prophylaxis prior to dental treatment
* Exhibiting gross oral pathology or a history of periodontal disease.
* Individuals with a history or are currently using birth control containing hormones.
* Individuals without a history (less than 1 year) of regular professional oral health care, including prophylaxis. (self-report)
* Pregnant, breastfeeding or planning for pregnancy within 3 months.
* Individuals who used antibiotics/chronically used NSAIDs
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Percent Composition of Human Gingival Tissue at Day 1 | Day 1
  Percentage of the human gingival biopsies that are epithelial, immune, or mesenchymal cells in health.
Percent Composition of Human Gingival Tissue at Day 21 | Day 21
  Percentage of the human gingival biopsies that are epithelial, immune, or mesenchymal cells during inflammation.
Percent Composition of Human Gingival Epithelial Cells at Day 1 | Day 1
  Percentage of the human gingival epithelial cell subtypes that are present (i.e. keratinocytes, Langerhans cells, etc.) in health.
Percent Composition of Human Gingival Epithelial Cells at Day 21 | Day 21
  Percentage of the human gingival epithelial cell subtypes that are present (i.e. keratinocytes, Langerhans cells, etc.) during inflammation.
Percent Composition of Human Gingival Immune Cells at Day 1 | Day 1
  Percentage of the human immune cell subtypes that are present (i.e. CD4, CD8, etc.) in health.
Percent Composition of Human Gingival Immune Cells at Day 21 | Day 21
  Percentage of the human immune cell subtypes that are present (i.e. CD4, CD8, etc.) during inflammation.
Percent Composition of Human Gingival Mesenchymal Cells at Day 1 | Day 1
  Percentage of the human mesenchymal cell subtypes that are present (i.e. stromal endothelial, etc.) in health.
Percent Composition of Human Gingival Mesenchymal Cells at Day 21 | Day 21
  Percentage of the human mesenchymal cell subtypes that are present (i.e. stromal endothelial, etc.) in health.
Genes Expressed In Epithelial Cells at Day 1 | Day 1
  Gene expression will be ranked by highest to lowest and a list of the top 100 genes in epithelial cells in health will be produced.
Genes Expressed In Epithelial Cells at Day 21 | Day 21
  Gene expression will be ranked by highest to lowest and a list of the top 100 genes in epithelial cells during inflammation will be produced.
Genes Expressed In Immune Cells at Day 1 | Day 1
  Gene expression will be ranked by highest to lowest and a list of the top 100 genes in immune cells in health will be produced.
Genes Expressed In Immune Cells at Day 21 | Day 21
  Gene expression will be ranked by highest to lowest and a list of the top 100 genes in immune cells during inflammation will be produced.
Genes Expressed In Mesenchymal Cells at Day 1 | Day 1
  Gene expression will be ranked by highest to lowest and a list of the top 100 genes in mesenchymal cells in health will be produced.
Genes Expressed In Mesenchymal Cells at Day 21 | Day 21
  Gene expression will be ranked by highest to lowest and a list of the top 100 genes in mesenchymal cells during inflammation will be produced.
Genes Expressed In Epithelial Cell Subtypes at Day 1 | Day 1
  Gene expression will be ranked by highest to lowest and a list of the top 100 genes in epithelial cell subtypes in health will be produced.
Genes Expressed In Epithelial Cell Subtypes at Day 21 | Day 21
  Gene expression will be ranked by highest to lowest and a list of the top 100 genes in epithelial cell subtypes during inflammation will be produced.
Genes Expressed In Immune Cell Subtypes at Day 1 | Day 1
  Gene expression will be ranked by highest to lowest and a list of the top 100 genes in immune cell subtypes in health will be produced.
Genes Expressed In Immune Cell Subtypes at Day 21 | Day 21
  Gene expression will be ranked by highest to lowest and a list of the top 100 genes in immune cell subtypes during inflammation will be produced.
Genes Expressed In Mesenchymal Cell Subtypes at Day 1 | Day 1
  Gene expression will be ranked by highest to lowest and a list of the top 100 genes in mesenchymal cell subtypes in health will be produced.
Genes Expressed In Mesenchymal Cell Subtypes at Day 21 | Day 21
  Gene expression will be ranked by highest to lowest and a list of the top 100 genes in mesenchymal cell subtypes during inflammation will be produced.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Byrd, DDS, PhD, Principal Investigator — Adams School of Dentistry, UNC Chapel Hill
Locations (1):
- Adams School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Single-cell RNA sequencing data will be shared through the Gene Expression Omnibus (GEO), a public functional genomics data repository supporting MIAME-compliant data submissions, which accepts sequence-based data. Gene list data will be searchable, cell by cell, through an online database. The files will be deposited both as raw reads (.fastq) and differential gene expression (.txt and .xlsx). Once data have been cleaned, assessed for differential gene expression, and validated by FISH/IHC, data will be made public. This will allow us to make this data freely available for others to investigate and reanalyze for their own purposes to accelerate further discoveries.
Time Frame: Gene expression data will be available for download once the manuscript has been accepted for publication.
Access Criteria: Gene expression lists by cell types will be provided to download freely in association with available journal access.